CLINICAL TRIAL: NCT03904420
Title: An Evidence Based Delivery Model of Care for Newly Implanted Adult CI Recipients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA determination of Fox software as class III medical device, not CDSS.
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAM5753
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Results first posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Sensorineural Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - New Model (Experimental): Standardized programming and testing method
  Interventions: Other: Clinical Education and Treatment Model
- Group B - Traditional Model (Active Comparator): Traditional clinical model which is not standardized across clinical sites
  Interventions: Other: Traditional Model

INTERVENTIONS:
Other: Clinical Education and Treatment Model — Patients will have self directed equipment education and standardized programming approaches
  Arms: Group A - New Model
Other: Traditional Model — Standard clinical practice and education
  Arms: Group B - Traditional Model

SUMMARY:
The clinical investigation is evaluating a new clinical model in a group of newly implanted subjects who have already been consented to CI surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are receiving a Nucleus® CI512, CI522, or CI532 electrodes
* 18 years and older
* Postlingual onset of hearing loss (onset of hearing loss >two years of age)
* Individuals who qualify for cochlear implantation using the clinics current CI candidacy criteria
* Individuals who have recently been implanted but not yet had their external device activated
* Willingness to participate in a study and comply with all study requirements
* Fluent in spoken English

Exclusion Criteria:

* Ossification or any other cochlear anomaly that might prevent insertion of less than 10 electrodes of the electrode array
* Diagnosis of retro-cochlear pathology
* Diagnosis of auditory neuropathy
* Subject considering an acoustic component in the implanted ear
* Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and use of the prosthetic device
* Unwillingness or inability to comply with all investigational requirements
* Severe-profound sensorineural hearing loss >30 years
* Previous cochlear implant in the contralateral ear. Additional cognitive, medical or social handicaps that would prevent completion of all study requirements as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Head and Neck Surgical Associates, Wichita Falls, Texas
  - Puget Sound ENT, Edmonds, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A - New Model | Group B - Traditional Model
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Study terminated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - New Model | Group B - Traditional Model | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Time Spent With Audiologist
Description: Change in the overall number of minutes of cochlear implant appointments over the first 6 months post activation in the new model (Group A) compared to the traditional model (Group B).
Time Frame: 6 months post activation
Population: No subjects completed all required visits and data for primary endpoints were not collected due to study termination shortly after execution commenced.
Arm/Group | Group A - New Model | Group B - Traditional Model
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Group A - New Model | Group B - Traditional Model
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PIs, no data was to be published prior to sponsor publishing. However, an agreement was in place with one site to provide presentation at upcoming conference for a poster presentation.

DOCUMENTS (2):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/20/NCT03904420/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03904420/SAP_001.pdf